CLINICAL TRIAL: NCT03890887
Title: Relative Bioavailability of a Single Oral Dose of BI 1291583 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects (an Open-label, Two-period, Fixed Sequence Study)
Brief Title: A Study in Healthy Men to Test How Itraconazole Influences the Amount of BI 1291583 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1397-0010; 2018-004214-17 (EudraCT Number)
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects: Reference followed by Test treatments (Experimental): Reference - BI 1291583 alone. Test - BI 1291583 + Itraconazole
  Interventions: Drug: BI 1291583; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 1291583 — Tablet
  Other Names: Verducatib
Drug: Itraconazole — Oral solution

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of BI 1291583 in plasma when given as oral single dose together with multiple oral doses of itraconazole (Test, T) as compared to when given alone as oral single dose (Reference, R).

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects with woman of childbearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of first administration of trial drug until 30 days after the last administration of trial drug administration
* Known relevant immunodeficiency
* Volunteers who have received live or live-attenuated vaccine in the 4 weeks prior to dosing
* Positive results for Hepatitis B antigen, Hepatitis C antibodies and/or human immunodeficiency virus (HIV) 1 antigen or HIV1/2 antibodies, at screening
* History and/or presence of tuberculosis; positive result for interferon gamma release assay (IGRA) (i.e., QuantiFERON TB-Gold)
* Subjects with signs of current gingivitis/periodontitis. Inspection of the oral cavity will be performed by the investigator
* Subjects with a history of hyperkeratosis or erythema in palms or soles.
* History of heart failure, or any evidence of ventricular dysfunction
* History of hereditary fructose intolerance
* History of drug-induced liver injury
* Liver enzymes (ALT, AST, GGT) above upper limit of normal at the screening examination
* Haemoglobin or red blood cell count below the lower limit of normal at the screening examination
* White blood cell count or neutrophil count outside the normal range at the screening examination

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 1291583 in plasma over the time interval from 0 to the last quantifiable data point | Up to 263 hours.
Maximum measured concentration of BI 1291583 in plasma | Up to 263 hours.

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity | Up to 263 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing